CLINICAL TRIAL: NCT00262847
Title: A Phase III Trial of Carboplatin and Paclitaxel Plus Placebo Versus Carboplatin and Paclitaxel Plus Concurrent Bevacizumab (NSC # 704865) Followed by Placebo, Versus Carboplatin and Paclitaxel Plus Concurrent and Extended Bevacizumab, in Women With Newly Diagnosed, Previously Untreated, Stage III or IV Epithelial Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Brief Title: Carboplatin and Paclitaxel With or Without Bevacizumab in Treating Patients With Stage III or Stage IV Ovarian Epithelial, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2009-00590; NCI-2009-00590 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000455114; GOG-0218 (Other: NRG Oncology); GOG-0218 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Results first posted 2013-09-18 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Malignant Ovarian Mixed Epithelial Tumor; Ovarian Brenner Tumor; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Adenocarcinoma; Ovarian Serous Adenocarcinoma; Ovarian Transitional Cell Carcinoma; Primary Peritoneal Serous Adenocarcinoma; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Primary Peritoneal Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Primary Peritoneal Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Primary Peritoneal Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Cancer; Stage IV Primary Peritoneal Cancer; Undifferentiated Fallopian Tube Carcinoma; Undifferentiated Ovarian Carcinoma
MeSH Terms: conditions — Brenner Tumor; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Carboplatin; Paclitaxel; Taxes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (placebo, paclitaxel, carboplatin) (Active Comparator): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Beginning in course 2, patients also receive placebo IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 6 courses. Beginning in course 7, patients receive placebo alone IV over 30-90 minutes on day 1. Treatment with placebo repeats every 21 days for up to 22 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Placebo; Other: Quality-of-Life Assessment
- Arm II (placebo, paclitaxel, carboplatin, bevacizumab) (Experimental): Patients receive paclitaxel and carboplatin as in arm I. Beginning in course 2, patients also receive bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 6 courses. Beginning in course 7, patients receive placebo alone IV over 30-90 minutes on day 1. Treatment with placebo repeats every 21 days for up to 22 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Placebo; Other: Quality-of-Life Assessment
- Arm III (paclitaxel, carboplatin, bevacizumab) (Experimental): Patients receive paclitaxel and carboplatin as in arm I. Beginning in course 2, patients also receive bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 6 courses. Beginning in course 7, patients receive bevacizumab alone IV over 30-90 minutes on day 1. Treatment with bevacizumab repeats every 21 days for up to 22 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
  Arms: Arm II (placebo, paclitaxel, carboplatin, bevacizumab); Arm III (paclitaxel, carboplatin, bevacizumab)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Placebo — Given IV
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm I (placebo, paclitaxel, carboplatin); Arm II (placebo, paclitaxel, carboplatin, bevacizumab)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial studies carboplatin, paclitaxel, and bevacizumab to see how well they work compared to carboplatin, paclitaxel, and placebo in treating patients with stage III or stage IV ovarian epithelial, primary peritoneal, or fallopian tube cancer. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. It is not yet known whether carboplatin, paclitaxel, and bevacizumab are more effective than carboplatin, paclitaxel, and placebo in treating ovarian epithelial, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the addition of 5 concurrent cycles of bevacizumab to 6 cycles of standard therapy (carboplatin and paclitaxel) (Arm II) increases the duration of progression-free survival (PFS) when compared to 6 cycles of standard therapy alone (Arm I) in women with newly diagnosed stage III (with any gross residual disease) and stage IV, epithelial ovarian, peritoneal primary or fallopian tube cancer.

II. To determine if the addition of 5 concurrent cycles of bevacizumab plus extended bevacizumab for 16 cycles beyond the 6 cycles of standard therapy (carboplatin and paclitaxel) (Arm III) increases progression-free survival when compared to 6 cycles of standard therapy (Arm I) in women with newly diagnosed stage III (with any gross residual disease) and stage IV, epithelial ovarian, peritoneal primary or fallopian tube cancer.

SECONDARY OBJECTIVES:

I. In the event that both Arm II and Arm III regimens are superior to the Arm I regimen with respect to progression-free survival, to determine whether the Arm III regimen prolongs progression-free survival when compared to the Arm II regimen.

II. To determine whether the Arm II or Arm III regimen increases the duration of overall survival when compared with the Arm I regimen.

III. To compare each of the experimental regimens to the Arm I regimen with respect to the incidence of severe toxicities or serious adverse events.

IV. To determine the impact on Quality of Life (QOL, as measured by the Functional Assessment of Cancer Therapy-Ovarian [FACT-O] trial outcome index [TOI]) following treatment with the above regimens.

TERTIARY OBJECTIVES:

I. To assess the relationship between angiogenic markers and clinical outcome including tumor response, progression-free survival and overall survival in patients randomized to standard cytotoxic chemotherapy (paclitaxel and carboplatin) without bevacizumab, with concurrent bevacizumab or with extended bevacizumab.

II. To assess the predictive value of a set of genes whose expression correlates with survival of patients with stage III (with any gross residual disease) and stage IV, epithelial ovarian, peritoneal primary or fallopian tube cancer.

III. To bank whole blood for research. IV. To determine if genetic variations in genes associated with essential hypertension including WNK lysine deficient protein kinase 1 (WNK1), G protein-coupled receptor kinase 4 (GRK4) and kallikrein B (KLKB1) predict which patients are likely to develop bevacizumab-induced hypertension.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30 minutes on day 1. Beginning in course 2, patients also receive placebo IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 6 courses. Beginning in course 7, patients receive placebo alone IV over 30-90 minutes on day 1. Treatment with placebo repeats every 21 days for up to 22 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive paclitaxel and carboplatin as in arm I. Beginning in course 2, patients also receive bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 6 courses. Beginning in course 7, patients receive placebo alone IV over 30-90 minutes on day 1. Treatment with placebo repeats every 21 days for up to 22 courses in the absence of disease progression or unacceptable toxicity.

ARM III: Patients receive paclitaxel and carboplatin as in arm I. Beginning in course 2, patients also receive bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 6 courses. Beginning in course 7, patients receive bevacizumab alone IV over 30-90 minutes on day 1. Treatment with bevacizumab repeats every 21 days for up to 22 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of epithelial ovarian cancer, peritoneal primary carcinoma or fallopian tube cancer; International Federation of Gynecology and Obstetrics (FIGO) stage III with any gross (macroscopic or palpable) residual disease or FIGO stage IV, defined surgically at the completion of initial abdominal surgery and with appropriate tissue available for histologic evaluation; the minimum surgery required was an abdominal surgery providing tissue for histologic evaluation and establishing and documenting the primary site and stage, as well as a maximal effort at tumor debulking; if additional surgery was performed, it should have been in accordance with appropriate surgery for ovarian or peritoneal carcinoma described in the Gynecologic Oncology Group (GOG) Surgical Procedures Manual; however, the surgeon is not required to have performed all of the items contained in this section of the GOG Surgical Procedures Manual; those patients with stage III cancer in which the largest maximal diameter of any residual tumor implant at the completion of this initial surgery is no greater than 1 cm will be defined as "optimal;" all others will be defined as "suboptimal;" measurable disease on post-operative imaging studies is not required for eligibility
* Patients with the following histologic epithelial cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma not otherwise specified (N.O.S.); however, the histologic features of the tumor must be compatible with a primary Müllerian epithelial adenocarcinoma; if doubt exists, it is recommended that the investigator should have the slides reviewed by an independent pathologist or, if necessary, the Pathology Co-Chair, prior to entry; patients may have co-existing fallopian tube carcinoma in-situ so long as the primary origin of invasive tumor is ovarian, peritoneal or fallopian tube
* Absolute neutrophil count (ANC) greater than or equal to 1,500/µl equivalent to Common Toxicity Criteria for Adverse Events version (v)3.0 (CTCAE) grade 1; this ANC cannot have been induced or supported by granulocyte colony stimulating factors
* Platelets greater than or equal to 100,000/µl; (CTCAE grade 0-1)
* Creatinine =< 1.5 x institutional upper limit normal (ULN), CTCAE grade 1
* Bilirubin less than or equal to 1.5 x ULN (CTCAE grade 1)
* Serum glutamic oxaloacetic transaminase (SGOT) and alkaline phosphatase less than or equal to 2.5 x ULN (CTCAE grade 1)
* Neuropathy (sensory and motor) less than or equal to CTCAE grade 1
* Prothrombin time (PT) such that international normalized ratio (INR) is =< 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin for management of venous thrombosis including pulmonary thrombo-embolus) and a partial thromboplastin time (PTT) < 1.2 times the upper limit of normal
* Patients with a GOG Performance Status of 0, 1, or 2
* Patients must be entered between 1 and 12 weeks after initial surgery performed for the combined purpose of diagnosis, staging and cytoreduction
* Patients with measurable and non-measurable disease are eligible; patients may or may not have cancer-related symptoms
* Patients who have met the pre-entry requirements
* An approved informed consent and authorization permitting release of personal health information must be signed by the patient or guardian
* Patients in this trial may receive ovarian estrogen +/- progestin replacement therapy as indicated at the lowest effective dose(s) for control of menopausal symptoms at any time, but not progestins for management of anorexia while on protocol directed therapy or prior to disease progression

Exclusion Criteria:

* Patients with a current diagnosis of borderline epithelial ovarian tumor (formerly "tumors of low malignant potential") or recurrent invasive epithelial ovarian, primary peritoneal or fallopian tube cancer treated with surgery only (such as patients with stage Ia or Ib low grade epithelial ovarian or fallopian tube cancers) are not eligible; patients with a prior diagnosis of a borderline tumor that was surgically resected and who subsequently develop an unrelated, new invasive epithelial ovarian, peritoneal primary or fallopian tube cancer are eligible, provided that they have not received prior chemotherapy for any ovarian tumor
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor including neo-adjuvant chemotherapy for their ovarian, primary peritoneal or fallopian tube cancer are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients who have received any targeted therapy (including but not limited to vaccines, antibodies, tyrosine kinase inhibitors) or hormonal therapy for management of their epithelial ovarian or peritoneal primary cancer
* Patients with synchronous primary endometrial cancer, or a past history of primary endometrial cancer, are excluded, unless all of the following conditions are met: stage not greater than I-B; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell or other FIGO grade 3 lesions
* With the exception of non-melanoma skin cancer and other specific malignancies as noted above, patients with other invasive malignancies who had (or have) any evidence of the other cancer present within the last five years or whose previous cancer treatment contraindicates this protocol therapy are excluded
* Patients with acute hepatitis or active infection that requires parenteral antibiotics
* Patients with serious non-healing wound, ulcer, or bone fracture; this includes history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days; patients with granulating incisions healing by secondary intention with no evidence of fascial dehiscence or infection are eligible but require weekly wound examinations
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of treatment on this study
* Patients with clinically significant cardiovascular disease; this includes:
* Uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 90 mm Hg
* Myocardial infarction or unstable angina < 6 months prior to registration
* New York Heart Association (NYHA) grade II or greater congestive heart failure
* Serious cardiac arrhythmia requiring medication; this does not include asymptomatic, atrial fibrillation with controlled ventricular rate
* CTCAE grade 2 or greater peripheral vascular disease (at least brief (< 24 hrs) episodes of ischemia managed non-surgically and without permanent deficit)
* History of CVA within six months
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* Patients with clinically significant proteinuria; urine protein should be screened by urine protein-creatinine ratio (UPCR); the UPCR has been found to correlate directly with the amount of protein excreted in a 24 hour urine collection; specifically, a UPCR of 1.0 is equivalent to 1.0 gram of protein in a 24 hour urine collection; obtain at least 4 ml of a random urine sample in a sterile container (does not have to be a 24 hour urine); send sample to lab with request for urine protein and creatinine levels [separate requests]; the lab will measure protein concentration (mg/dL) and creatinine concentration (mg/dL); the UPCR is derived as follows: protein concentration (mg/dL)/creatinine (mg/dL); patients must have a UPCR < 1.0 to allow participation in the study
* Patients with or with anticipation of invasive procedures as defined below:
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to the first date of bevacizumab/placebo therapy (cycle 2)
* Major surgical procedure anticipated during the course of the study; this includes, but is not limited to abdominal surgery (laparotomy or laparoscopy) prior to disease progression, such as colostomy or enterostomy reversal, interval or secondary cytoreductive surgery, or second look surgery; please consult with the study chair prior to patient entry for any questions related to the classification of surgical procedures
* Core biopsy, within 7 days prior to the first date of bevacizumab/placebo therapy (cycle 2)
* Patients with GOG Performance Grade of 3 or 4
* Patients who are pregnant or nursing; bevacizumab should not be administered to nursing women; patients of childbearing potential must agree to use contraceptive measures during study therapy and for at least six months after completion of bevacizumab therapy
* Patients who have received prior therapy with any anti-vascular endothelial growth factor (VEGF) drug, including bevacizumab
* Patients with clinical symptoms or signs of gastrointestinal obstruction and who require parenteral hydration and/or nutrition
* Patients with medical history or conditions not otherwise previously specified which in the opinion of the investigator should exclude participation in this study; the investigator should feel free to consult the study chair or study co-chairs for uncertainty in this regard

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1873 (Actual)
Dates: Start 2005-09; Primary Completion 2010-11 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Burger, Principal Investigator — NRG Oncology
Locations (631):
- United States (613):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Banner Thunderbird Medical Center, Glendale, Arizona
  - Banner Desert Medical Center, Mesa, Arizona
  - Banner Baywood Medical Center, Mesa, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Western Regional CCOP, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Highlands Oncology Group PA - Fayetteville, Fayetteville, Arkansas
  - Washington Regional Medical Center - Fayetteville, Fayetteville, Arkansas
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Northbay Cancer Center, Fairfield, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Cancer Care Associates of Fresno Medical Group Inc, Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute, Palo Alto, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Cancer Center of Santa Barbara, Santa Barbara, California
  - Santa Barbara Hematology Oncology Group Inc-Santa Barbara, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Colorado Gynecologic Oncology Group, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Rocky Mountain Gynecologic Oncology PC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Saint Vincent's Medical Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Bayfront Outpatient Health Clinic, St. Petersburg, Florida
  - Florida Cancer Specialists-West Palm Beach, West Palm Beach, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Grady Health System, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Georgia Regents University Medical Center, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Hospital, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Chicago Gynecologic Oncology SC, Palatine, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Franciscan St. Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium CCOP, South Bend, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, Waterloo, Iowa
  - Covenant Medical Center, Waterloo, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Shawnee Mission Medical Center-KCCC, Shawnee Mission, Kansas
  - Stormont-Vail Regional Health Center, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Christus Schumpert Saint Mary's Place, Shreveport, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Memorial Hospital at Easton - Shore Regional Cancer Center, Easton, Maryland
  - The Memorial Hospital at Easton, Easton, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Associates in Oncology Hematology PC -Kensington, Kensington, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Kaiser Permanente - Towson Medical Center, Lutherville, Maryland
  - Kaiser Permanente - Shady Grove Medical Center, Rockville, Maryland
  - Maryland Oncology Hematology PA-Aquilino Cancer Center, Rockville, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Berkshire Hematology Oncology PC, Pittsfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Commonwealth Hematology Oncology PC-Worcester, Worcester, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Spectrum Health-Blodgett Campus, Grand Rapids, Michigan
  - Gynecologic Oncology of West Michigan PLLC, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - McLaren-Northern Michigan, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Providence Hospital-Southfield Cancer Center, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Hubert H Humphrey Cancer Center, Robbinsdale, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota NCI Community Oncology Research Program, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Regional Medical Center, Jefferson City, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Medical Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Exeter Hospital, Exeter, New Hampshire
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Frisbie Hospital, Rochester, New Hampshire
  - Ocean Medical Center, Brick, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical CCOP, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Northern New Jersey CCOP, Hackensack, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - UMDNJ - New Jersey Medical School, Newark, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Island Gynecologic Oncology, Brightwaters, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Queens Hospital Center, Jamaica, New York
  - North Shore University Hospital, Manhasset, New York
  - Orange Regional Medical Center, Middletown, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - North Shore-LIJ Health System/Center for Advanced Medicine, New Hyde Park, New York
  - Laura and Issac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Saint Joseph's Hospital Health Center, Syracuse, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Good Samaritan Hospital Medical Center, West Islip, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Gynecologic Oncology Network, Greenville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Southeast Cancer Consortium-Upstate NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates-Midtown, Tulsa, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Kaiser Permanente, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Chestnut Hill Health System, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Mainline Health CCOP, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Hospital, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Chattanooga Gynecological Oncology, Chattanooga, Tennessee
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - East Tennessee State University, Johnson City, Tennessee
  - Knoxville Gynecologic Cancer Specialists PC, Knoxville, Tennessee
  - University of Tennesee Health Science Center, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Northern Virginia Pelvic Surgery Associates, Annandale, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Kaiser Permanente - Fair Oaks Medical Center, Fairfax, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Rappahannock General Hospital, Kilmarnock, Virginia
  - Bon Secours Mary Immaculate Hospital, Newport News, Virginia
  - Virginia Oncology Associates - Lake Wright, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Virginia Mason CCOP, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest CCOP, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Medical Consultants Limited, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic - Slinger, Slinger, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming
- Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
- Japan (10):
  - Tohoku University School of Medicine, Sendai, Aoba-ku
  - Kure National Hospital, Kure, Hiroshima
  - Iwate Medical University School of Medicine, Morioka, Iwate
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - Keio University, Shinjuku-ku, Tokyo
  - National Hospital Organization-Kobe Medical Center, Kobe
  - Shikoku Cancer Center, Matsuyama
  - Saitama Medical University International Medical Center, Saitama
  - National Cancer Center Hospital, Tokyo
  - Tottori University, Tottori
- South Korea (7):
  - Samsung Medical Center, Seoul, Korea
  - Seoul National University Hospital, Seoul
  - Yongdong Severence Hospital, Seoul
  - Asan Medical Center, Seoul
  - Korea Cancer Center Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Kangnam Sacred Heart Hospital, Youngdungpo-gu

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] You B, Purdy C, Copeland LJ, Swisher EM, Bookman MA, Fleming G, Coleman R, Randall LM, Tewari KS, Monk BJ, Mannel RS, Walker JL, Cappuccini F, Cohn D, Muzaffar M, Mutch D, Wahner-Hendrickson A, Martin L, Colomban O, Burger RA. Identification of Patients With Ovarian Cancer Experiencing the Highest Benefit From Bevacizumab in the First-Line Setting on the Basis of Their Tumor-Intrinsic Chemosensitivity (KELIM): The GOG-0218 Validation Study. J Clin Oncol. 2022 Dec 1;40(34):3965-3974. doi: 10.1200/JCO.22.01207. Epub 2022 Oct 17. PMID 36252167
- [Derived] Morgan RD, Ferreras C, Peset I, Avizienyte E, Renehan AG, Edmondson RJ, Murphy AD, Nicum S, Van Brussel T, Clamp AR, Lambrechts D, Zhou C, Jayson GC. c-MET/VEGFR-2 co-localisation impacts on survival following bevacizumab therapy in epithelial ovarian cancer: an exploratory biomarker study of the phase 3 ICON7 trial. BMC Med. 2022 Feb 11;20(1):59. doi: 10.1186/s12916-022-02270-y. PMID 35144591
- [Derived] Tewari KS, Burger RA, Enserro D, Norquist BM, Swisher EM, Brady MF, Bookman MA, Fleming GF, Huang H, Homesley HD, Fowler JM, Greer BE, Boente M, Liang SX, Ye C, Bais C, Randall LM, Chan JK, Ferriss JS, Coleman RL, Aghajanian C, Herzog TJ, DiSaia PJ, Copeland LJ, Mannel RS, Birrer MJ, Monk BJ. Final Overall Survival of a Randomized Trial of Bevacizumab for Primary Treatment of Ovarian Cancer. J Clin Oncol. 2019 Sep 10;37(26):2317-2328. doi: 10.1200/JCO.19.01009. Epub 2019 Jun 19. PMID 31216226
- [Derived] Eskander RN, Kauderer J, Tewari KS, Mannel RS, Bristow RE, O'Malley DM, Rubin SC, Glaser GE, Hamilton CA, Fujiwara K, Huh WK, Ueland F, Stephan JM, Burger RA. Correlation between Surgeon's assessment and radiographic evaluation of residual disease in women with advanced stage ovarian cancer reported to have undergone optimal surgical cytoreduction: An NRG Oncology/Gynecologic Oncology Group study. Gynecol Oncol. 2018 Jun;149(3):525-530. doi: 10.1016/j.ygyno.2018.03.043. Epub 2018 Mar 15. PMID 29550184
- [Derived] Tewari KS, Java JJ, Eskander RN, Monk BJ, Burger RA. Early initiation of chemotherapy following complete resection of advanced ovarian cancer associated with improved survival: NRG Oncology/Gynecologic Oncology Group study. Ann Oncol. 2016 Jan;27(1):114-21. doi: 10.1093/annonc/mdv500. Epub 2015 Oct 20. PMID 26487588
- [Derived] Monk BJ, Huang HQ, Burger RA, Mannel RS, Homesley HD, Fowler J, Greer BE, Boente M, Liang SX, Wenzel L. Patient reported outcomes of a randomized, placebo-controlled trial of bevacizumab in the front-line treatment of ovarian cancer: a Gynecologic Oncology Group Study. Gynecol Oncol. 2013 Mar;128(3):573-8. doi: 10.1016/j.ygyno.2012.11.038. Epub 2012 Dec 4. PMID 23219660
- [Derived] Burger RA, Brady MF, Bookman MA, Fleming GF, Monk BJ, Huang H, Mannel RS, Homesley HD, Fowler J, Greer BE, Boente M, Birrer MJ, Liang SX; Gynecologic Oncology Group. Incorporation of bevacizumab in the primary treatment of ovarian cancer. N Engl J Med. 2011 Dec 29;365(26):2473-83. doi: 10.1056/NEJMoa1104390. PMID 22204724
- [Derived] Vaughan S, Coward JI, Bast RC Jr, Berchuck A, Berek JS, Brenton JD, Coukos G, Crum CC, Drapkin R, Etemadmoghadam D, Friedlander M, Gabra H, Kaye SB, Lord CJ, Lengyel E, Levine DA, McNeish IA, Menon U, Mills GB, Nephew KP, Oza AM, Sood AK, Stronach EA, Walczak H, Bowtell DD, Balkwill FR. Rethinking ovarian cancer: recommendations for improving outcomes. Nat Rev Cancer. 2011 Sep 23;11(10):719-25. doi: 10.1038/nrc3144. PMID 21941283

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2005 and June 2009, 1873 women were enrolled from 336 institutions in the United States, Canada, South Korea, and Japan.
Groups:
- Arm I (Placebo, Paclitaxel, Carboplatin): Control therapy:
  Cycles 1-6 received paclitaxel, 175 mg/m2 plus carboplatin AUC 6 plus placebo (starting in cycle 2) every 3 weeks.
  Cycles 7-22 received placebo every 3 weeks.
- Arm II (Placebo, Paclitaxel, Carboplatin, Bevacizumab): Bevacizumab-initiation therapy:
  Cycles 1-6 received paclitaxel, 175 mg/m2 plus carboplatin AUC 6 plus bevacizumab, 15 mg/kg (starting in cycle 2) every 3 weeks.
  Cycles 7-22 received placebo every 3 weeks.
- Arm III (Paclitaxel, Carboplatin, Bevacizumab): Bevacizumab-throughout therapy:
  Cycles 1-6 received paclitaxel, 175 mg/m2 plus carboplatin AUC 6 plus bevacizumab, 15 mg/kg (starting in cycle 2) every 3 weeks.
  Cycles 7-22 received bevacizumab, 15 mg/kg every 3 weeks.
Period: Overall Study
Arm/Group | Arm I (Placebo, Paclitaxel, Carboplatin) | Arm II (Placebo, Paclitaxel, Carboplatin, Bevacizumab) | Arm III (Paclitaxel, Carboplatin, Bevacizumab)
Started | 625 (Total enrolled and included in efficacy analysis) | 625 (Total enrolled and included in efficacy analysis) | 623 (Total enrolled and included in efficacy analysis)
Completed | 107 | 112 | 227
Not Completed | 518 | 513 | 396
Not completed — Disease Progression | 309 | 274 | 195
Not completed — Patient Refusal | 41 | 52 | 47
Not completed — Adverse Event | 74 | 88 | 108
Not completed — Death | 8 | 8 | 11
Not completed — Concomitant disease | 3 | 2 | 4
Not completed — Other Reasons | 79 | 88 | 27
Not completed — Did not receive study treatment | 4 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Placebo, Paclitaxel, Carboplatin) | Arm II (Placebo, Paclitaxel, Carboplatin, Bevacizumab) | Arm III (Paclitaxel, Carboplatin, Bevacizumab) | Total
Number analyzed (Participants) | 625 | 625 | 623 | 1873
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (10.9) | 60.1 (10.3) | 59.7 (10.6) | 59.7 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 625 | 625 | 623 | 1873
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participant]
  Non-Hispanic white | 526 | 519 | 521 | 1566
  Asian | 41 | 37 | 39 | 117
  Non-Hispanic black | 25 | 28 | 27 | 80
  Hispanic | 21 | 28 | 25 | 74
  Other or unspecified | 12 | 13 | 11 | 36
Region of Enrollment [Number; unit: participants]
  United States | 596 | 596 | 599 | 1791
  Canada | 1 | 5 | 3 | 9
  Japan | 21 | 12 | 12 | 45
  Korea, Republic of | 7 | 12 | 9 | 28
Gynecologic Oncology Group (GOG) Performance Status [Number; unit: participants] — 5-point, ordinal scale specifying patient's ability to perform activities from 0(fully active) to 4(completely disabled, no self-care).
  participants
    0 - fully active | 311 | 315 | 305 | 931
    1 - restricted strenuous activity, ambulatory | 272 | 270 | 267 | 809
    2 - ambulatory, difficulty walking | 42 | 40 | 51 | 133
    3 - limited self-care, partly confined to bed | 0 | 0 | 0 | 0
    4 - completely disabled, no self-care | 0 | 0 | 0 | 0
International Federation of Gynecologic and Obstetrics (FIGO) Stage [Number; unit: participants] — Clinical staging for primary carcinoma of the ovary (1985) from Stage 1 (limited to ovaries) to Stage 4 (distant metastatis)
  participants
    1-limited to ovaries | 0 | 0 | 0 | 0
    1A-1 ovary involved, no ascites | 0 | 0 | 0 | 0
    1B-both ovaries involved, no ascites | 0 | 0 | 0 | 0
    1C-disease with capsules ruptured or ascites | 0 | 0 | 0 | 0
    2-disease with pelvic extension | 0 | 0 | 0 | 0
    2A-disease with extension to uterus and or tubes | 0 | 0 | 0 | 0
    2B-disease with extension to other pelvic tissues | 0 | 0 | 0 | 0
    2C-disease with capsules ruptured or ascites | 0 | 0 | 0 | 0
    3-disease w/ macroscopic implants outside pelvis | 218 | 205 | 216 | 639
    3-disease w/ implants > 1 cm outside pelvis | 254 | 256 | 242 | 752
    3A-disease w/ microscopic implants, negative nodes | 0 | 0 | 0 | 0
    3B-disease w/ abdominal implants <2cm, neg nodes | 0 | 0 | 0 | 0
    3C-disease w/ abdominal implants >2cm, pos nodes | 0 | 0 | 0 | 0
    4-distant metastatis | 153 | 164 | 165 | 482
Histologic Type [Number; unit: participants] — Histologic(cell) type was obtained from the central GOG Pathology Committee review updated in September 2010.
  participants
    Serous adenocarcinoma | 541 | 519 | 524 | 1584
    Endometrioid | 21 | 14 | 24 | 59
    Clear cell | 12 | 23 | 20 | 55
    Mucinous | 6 | 5 | 8 | 19
    Other or not specified | 45 | 64 | 47 | 156
Tumor Grade [Number; unit: participants] — Tumor grade was obtained from the central GOG Pathology Committee review updated in September 2010. All clear-cell tumors were classified as grade 3.
  participants
    3 | 445 | 465 | 460 | 1370
    2 | 102 | 86 | 97 | 285
    1 | 36 | 28 | 18 | 82
    Not graded | 42 | 46 | 48 | 136

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Median progression-free survival (PFS). Onset of progression could be based on radiographic (RECIST) criteria or rising CA-125 (GCIG criteria).
Time Frame: From study entry until first disease progression, death or date of last contact, up to 6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Placebo, Paclitaxel, Carboplatin) | Arm II (Placebo, Paclitaxel, Carboplatin, Bevacizumab) | Arm III (Paclitaxel, Carboplatin, Bevacizumab)
Number analyzed (Participants) | 625 | 625 | 623
months | 11.0 [10.2 to 12.0] | 12.3 [11.4 to 12.8] | 15.3 [14.2 to 16.1]
Statistical Analysis 1: Comparison: Arm I (Placebo, Paclitaxel, Carboplatin) vs Arm II (Placebo, Paclitaxel, Carboplatin, Bevacizumab); Test type: Superiority or Other; p = 0.448, Regression, Cox; Proportional Hazards model stratified by stage of disease and size of residual disease following initial staging surgery; Hazard Ratio (HR) = 0.954, 95% CI [0.844 to 1.078]
Statistical Analysis 2: Comparison: Arm I (Placebo, Paclitaxel, Carboplatin) vs Arm III (Paclitaxel, Carboplatin, Bevacizumab); Test type: Superiority or Other; p < 0.001, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.765, 95% CI [0.676 to 0.866]

2. Secondary Outcome: Overall Survival
Description: Median overall survival (OS)
Time Frame: From study entry to death or last contact, up to 6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Placebo, Paclitaxel, Carboplatin) | Arm II (Placebo, Paclitaxel, Carboplatin, Bevacizumab) | Arm III (Paclitaxel, Carboplatin, Bevacizumab)
Number analyzed (Participants) | 625 | 625 | 623
months | 40.6 [37.1 to 45.5] | 38.7 [35.2 to 42.1] | 43.8 [39.7 to 49.0]
Statistical Analysis 1: Comparison: Arm I (Placebo, Paclitaxel, Carboplatin) vs Arm II (Placebo, Paclitaxel, Carboplatin, Bevacizumab); Test type: Superiority or Other; p = 0.410, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.069, 95% CI [0.912 to 1.255]
Statistical Analysis 2: Comparison: Arm I (Placebo, Paclitaxel, Carboplatin) vs Arm III (Paclitaxel, Carboplatin, Bevacizumab); Test type: Superiority or Other; p = 0.131, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.880, 95% CI [0.746 to 1.039]

3. Secondary Outcome: Frequency and Severity (Grade 3 or Above) of Adverse Events Assessed by Common Terminology Criteria for Adverse Events Version 3.0
Description: Eligible and Evaluable patients
Time Frame: Up to 5 years
Population: Eligible and evaluable patients
Measure: Count of Participants; unit: Participants
Groups:
- Arm I Toxicities (Placebo, Paclitaxel, Carboplatin): Control therapy:
  Cycles 1-6 received paclitaxel, 175 mg/m2 plus carboplatin AUC 6 plus placebo (starting in cycle 2) every 3 weeks.
  Cycles 7-22 received placebo every 3 weeks.
- Arm II Toxicities (Placabo,Paclitaxel,Carboplatin,Bevacizumab): Bevacizumab-initiation therapy:
  Cycles 1-6 received paclitaxel, 175 mg/m2 plus carboplatin AUC 6 plus bevacizumab, 15 mg/kg (starting in cycle 2) every 3 weeks.
  Cycles 7-22 received placebo every 3 weeks.
- Arm III Toxicities (Paclitaxel, Carboplatin, Bevacizumab): Bevacizumab-throughout therapy:
  Cycles 1-6 received paclitaxel, 175 mg/m2 plus carboplatin AUC 6 plus bevacizumab, 15 mg/kg (starting in cycle 2) every 3 weeks.
  Cycles 7-22 received bevacizumab, 15 mg/kg every 3 weeks.
Arm/Group | Arm I Toxicities (Placebo, Paclitaxel, Carboplatin) | Arm II Toxicities (Placabo,Paclitaxel,Carboplatin,Bevacizumab) | Arm III Toxicities (Paclitaxel, Carboplatin, Bevacizumab)
Number analyzed (Participants) | 621 | 624 | 619
Participants
  White blood cell | 317 | 328 | 327
  Absolute neutrophil count | 540 | 543 | 536
  Hemoglobin | 91 | 86 | 74
  Platelets | 93 | 122 | 131
  Other hematologic | 13 | 13 | 9
  Allergy/Immunology | 23 | 25 | 14
  Auditory/Ear | 1 | 1 | 2
  hypertension | 10 | 36 | 65
  Cardiac | 14 | 12 | 18
  Coagulation | 5 | 7 | 8
  Constitutional | 62 | 61 | 83
  Dermatologic | 13 | 20 | 16
  Endocrine | 4 | 4 | 2
  Gastrointestinal | 96 | 112 | 122
  Genitourinary/Renal | 13 | 8 | 8
  Hemorrhage | 5 | 9 | 15
  Hepatobiliary | 2 | 1 | 3
  Infection | 75 | 73 | 95
  Lymphatics | 4 | 3 | 3
  Metabolic | 91 | 87 | 101
  Musculoskeletal | 16 | 17 | 21
  Neurosensory | 23 | 26 | 28
  Other neurological | 44 | 42 | 65
  Ocular/Visual | 4 | 1 | 4
  Pain | 74 | 82 | 101
  Pulmonary | 29 | 36 | 32
  Vascular | 37 | 33 | 40
  Death, not CTC coded | 5 | 8 | 10
  Sexual/Reproductive | 1 | 0 | 0

4. Secondary Outcome: Impact on Quality of Life Measured by the Functional Assessment of Cancer Therapy-Ovary Trial Outcome Index (FACT-O TOI)
Description: Estimated least squares means from a mixed module of Quality of Life (QOL) scores at each assessment point, adjusted for baseline score and patient's age. Note: The range of possible scores of the FACT-O TOI is 0 - 104 for all treatment groups and at all visits. A higher score indicates better QOL. Baseline mean scores are raw means.
Time Frame: At baseline, 9, 18, 36, 60, and 84 weeks
Population: Number of valid QOL assessments do not total number of patients randomized in study.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Placebo, Paclitaxel, Carboplatin) | Arm II (Placebo, Paclitaxel, Carboplatin, Bevacizumab) | Arm III (Paclitaxel, Carboplatin, Bevacizumab)
Number analyzed (Participants) | 625 | 625 | 623
units on a scale
  prior to treatment | 68.2 (0.64) | 68.0 (0.66) | 67.4 (0.65)
  prior to cycle 4 | 73.8 (0.53) | 71.1 (0.56) | 70.9 (0.54)
  prior to cycle 7 | 76.0 (0.54) | 74.3 (0.56) | 73.8 (0.58)
  prior to cycle 13 | 80.6 (0.62) | 80.5 (0.62) | 79.9 (0.58)
  prior to cycle 21 | 77.6 (0.73) | 79.1 (0.71) | 78.6 (0.66)
  6 months followup | 75.8 (0.78) | 77.6 (0.75) | 77.8 (0.75)

ADVERSE EVENTS:
Time Frame: All Adverse Events(AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adeverse Events (SAEs) considered to be treatment related for up to 5 years after stopping study treatment.
Arm/Group | Arm I (Placebo, Paclitaxel, Carboplatin) | Arm II (Placebo, Paclitaxel, Carboplatin, Bevacizumab) | Arm III (Paclitaxel, Carboplatin, Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 239/621 | 257/624 | 287/619
Other Adverse Events (participants affected / at risk) | 589/621 | 593/624 | 588/619
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Placebo, Paclitaxel, Carboplatin) (N=621) | Arm II (Placebo, Paclitaxel, Carboplatin, Bevacizumab) (N=624) | Arm III (Paclitaxel, Carboplatin, Bevacizumab) (N=619)
Allergy/Immunology - Other (Immune system disorders) | 0 | 0 | 1
Allergic Reaction/Hypersensitivity (Immune system disorders) | 3 | 6 | 4
Myelodysplasia (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutrophils (Blood and lymphatic system disorders) | 14 | 15 | 13
Platelets (Blood and lymphatic system disorders) | 1 | 2 | 0
Leukocytes (Blood and lymphatic system disorders) | 1 | 2 | 3
Hemoglobin (Blood and lymphatic system disorders) | 3 | 2 | 1
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 3 | 0 | 1
Cardiac Arrhythmia - Other (Cardiac disorders) | 1 | 0 | 0
S/N Arrhythmia: Atrial Flutter (Cardiac disorders) | 1 | 0 | 0
Vasovagal Episode (Cardiac disorders) | 0 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 2
S/N Arrhythmia:supraventricular Nos (Cardiac disorders) | 0 | 1 | 0
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac Ischemia/Infarction (Cardiac disorders) | 2 | 2 | 1
Hypertension (Cardiac disorders) | 0 | 4 | 5
Left Venticular Diastolic Dysfunction (Cardiac disorders) | 0 | 0 | 1
Cardiac General - Other (Cardiac disorders) | 0 | 1 | 0
Cardiac Troponin I (Ctni) (Cardiac disorders) | 0 | 1 | 0
Hypotension (Cardiac disorders) | 1 | 0 | 2
Inr (Vascular disorders) | 0 | 0 | 1
Fever (General disorders) | 3 | 2 | 5
Fatigue (General disorders) | 1 | 4 | 2
Death No Ctcae Term - Disease Progression Nos (General disorders) | 0 | 4 | 1
Death No Ctcae Term - Death Nos (General disorders) | 0 | 0 | 2
Death No Ctcae Term - Multi-Organ Failure (General disorders) | 1 | 0 | 0
Death No Ctcae Term - Sudden Death (General disorders) | 1 | 2 | 2
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 3 | 4 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Endocrine - Other (Endocrine disorders) | 0 | 0 | 1
Fistula, Gi - Colon/Cecum/Appendix (Gastrointestinal disorders) | 1 | 2 | 1
Obstruction, Gi - Ileum (Gastrointestinal disorders) | 0 | 0 | 1
Necrosis, Gi - Small Bowel Nos (Gastrointestinal disorders) | 0 | 1 | 0
Perforation, Gi - Colon (Gastrointestinal disorders) | 0 | 4 | 4
Fistula, Gi - Ileum (Gastrointestinal disorders) | 1 | 0 | 0
Fistula, Gi - Small Bowel Nos (Gastrointestinal disorders) | 0 | 2 | 1
Fistula, Gi - Rectum (Gastrointestinal disorders) | 1 | 1 | 1
Obstruction, Gi - Colon (Gastrointestinal disorders) | 2 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis (Functional/Sympt) - Esophagus (Gastrointestinal disorders) | 0 | 0 | 1
Leak, Gi - Large Bowel (Gastrointestinal disorders) | 0 | 0 | 1
Perforation, Gi - Rectum (Gastrointestinal disorders) | 1 | 0 | 0
Leak, Gi - Rectum (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 5 | 8 | 3
Fistula, Gi - Abdomen Nos (Gastrointestinal disorders) | 0 | 0 | 1
Obstruction, Gi - Duodenal (Gastrointestinal disorders) | 0 | 1 | 0
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 13 | 13 | 15
Colitis (Gastrointestinal disorders) | 3 | 1 | 5
Obstruction, Gi - Jejunum (Gastrointestinal disorders) | 0 | 1 | 0
Perforation, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 12 | 9 | 6
Anorexia (Gastrointestinal disorders) | 2 | 0 | 0
Dehydration (Gastrointestinal disorders) | 9 | 10 | 11
Constipation (Gastrointestinal disorders) | 4 | 4 | 3
Nausea (Gastrointestinal disorders) | 4 | 3 | 5
Gastrointestinal - Other (Gastrointestinal disorders) | 1 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 3 | 7
Prolapse Of Stoma, Gi (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhage, Gu - Vagina (Vascular disorders) | 0 | 0 | 1
Hemorrhage, Gi - Rectum (Vascular disorders) | 1 | 0 | 0
Hemorrhage, Gi - Upper Gi Nos (Vascular disorders) | 0 | 1 | 0
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 0 | 0 | 1
Hematoma (Vascular disorders) | 1 | 0 | 0
Hemorrhage, Gi - Lower Gi Nos (Vascular disorders) | 0 | 0 | 2
Hemorrhage, Gu - Kidney (Vascular disorders) | 0 | 0 | 1
Hemorrhage, Gi - Stomach (Vascular disorders) | 0 | 1 | 1
Hemorrhage, Cns (Vascular disorders) | 0 | 0 | 1
Hemorrhage/Bleeding - Other (Vascular disorders) | 0 | 0 | 1
Hepatobiliary/Pancreas - Other (Hepatobiliary disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 3
Pancreatitis (Hepatobiliary disorders) | 1 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Wound (Infections and infestations) | 1 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 3 | 1 | 1
Inf W/Gr 3 Or 4 Anc: Salivary Gland (Infections and infestations) | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Skin (Cellulitis) (Infections and infestations) | 1 | 0 | 1
Inf W/Gr 3 Or 4 Anc: External Ear (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 2 | 3 | 3
Inf W/Gr 3 Or 4 Anc: Peritoneal Cavity (Infections and infestations) | 0 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Esophagus (Infections and infestations) | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bone (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 3 | 3 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 1 | 2 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 2 | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Catheter-Related (Infections and infestations) | 1 | 2 | 2
Febrile Neutropenia (Infections and infestations) | 16 | 20 | 21
Inf W/Nml Or Gr 1 Or 2 Anc: Rectum (Infections and infestations) | 0 | 1 | 0
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 0 | 1 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 1 | 3 | 4
Infection - Other (Infections and infestations) | 4 | 4 | 3
Inf W/Gr 3 Or 4 Anc: Bladder (Urinary) (Infections and infestations) | 0 | 2 | 3
Opportunisitic Inf Assoc. W/Gr 2 Lymphopenia (Infections and infestations) | 1 | 0 | 0
Colitis, Infectious (Eg.C. Difficile) (Infections and infestations) | 1 | 3 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 1 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Abdomen Nos (Infections and infestations) | 3 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Pelvis Nos (Infections and infestations) | 0 | 1 | 0
Inf Unknown Anc: Neck Nos (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc:peritoneal Cavity (Infections and infestations) | 1 | 0 | 1
Inf Unknown Anc: Catheter-Related (Infections and infestations) | 0 | 2 | 0
Inf W/Gr 3 Or 4 Anc: Pelvis Nos (Infections and infestations) | 0 | 2 | 0
Inf W/Gr 3 Or 4 Anc: Upper Airway Nos (Infections and infestations) | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Sinus (Infections and infestations) | 1 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Lung (Pneumonia) (Infections and infestations) | 3 | 2 | 1
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 3 | 4 | 3
Inf W/Gr 3 Or 4 Anc: Catheter-Related (Infections and infestations) | 2 | 0 | 1
Lymphocele (Blood and lymphatic system disorders) | 1 | 0 | 1
Proteinuria (Metabolism and nutrition disorders) | 0 | 0 | 1
Creatinine (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Alt (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Soft Tissue Necrosis - Abdomen (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint-Function (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 5 | 4 | 2
Psychosis (Nervous system disorders) | 1 | 1 | 0
Neurology - Other (Nervous system disorders) | 1 | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 1 | 1
Mood Alteration - Depression (Nervous system disorders) | 1 | 0 | 1
Mood Alteration - Anxiety (Nervous system disorders) | 0 | 1 | 1
Seizure (Nervous system disorders) | 1 | 0 | 1
Cognitive Disturbance (Nervous system disorders) | 0 | 2 | 0
Cns Ischemia (Nervous system disorders) | 3 | 0 | 5
Confusion (Nervous system disorders) | 1 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 2
Neuropathy-Sensory (Nervous system disorders) | 2 | 0 | 0
Neuropathy-Motor (Nervous system disorders) | 0 | 2 | 1
Cataract (Eye disorders) | 0 | 0 | 2
Pain - Other (General disorders) | 0 | 1 | 1
Pain: Pelvis (General disorders) | 0 | 1 | 1
Pain: Chest /Thorax Nos (General disorders) | 1 | 1 | 4
Pain: Chest Wall (General disorders) | 0 | 1 | 0
Pain: Pleura (General disorders) | 0 | 1 | 0
Pain: Head/Headache (General disorders) | 1 | 1 | 0
Pain: Intestine (General disorders) | 1 | 0 | 0
Pain: Back (General disorders) | 0 | 1 | 1
Pain: Joint (General disorders) | 1 | 0 | 0
Pain: Bone (General disorders) | 0 | 0 | 1
Pain: Kidney (General disorders) | 1 | 0 | 0
Pain: Pain Nos (General disorders) | 1 | 0 | 0
Pain: Rectum (General disorders) | 2 | 1 | 0
Pain: Abdominal Pain Nos (General disorders) | 8 | 8 | 12
Pain: Muscle (General disorders) | 0 | 0 | 1
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 7
Perforation, Gu - Vagina (Renal and urinary disorders) | 1 | 0 | 0
Obstruction, Gu - Ureter (Renal and urinary disorders) | 0 | 1 | 0
Fistula, Gu - Vagina (Renal and urinary disorders) | 1 | 0 | 0
2nd Mal: Poss. Related To Cancer Rx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Artery Injury - Carotid (Vascular disorders) | 0 | 1 | 0
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 2 | 5 | 2
Thrombosis/Thrombus/Embolism (Vascular disorders) | 17 | 14 | 21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Placebo, Paclitaxel, Carboplatin) (N=621) | Arm II (Placebo, Paclitaxel, Carboplatin, Bevacizumab) (N=624) | Arm III (Paclitaxel, Carboplatin, Bevacizumab) (N=619)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 56 | 65 | 68
Rhinitis (Immune system disorders) | 67 | 93 | 98
Tinnitus (Ear and labyrinth disorders) | 28 | 18 | 32
Neutrophils (Blood and lymphatic system disorders) | 589 | 591 | 588
Platelets (Blood and lymphatic system disorders) | 419 | 426 | 435
Leukocytes (Blood and lymphatic system disorders) | 578 | 593 | 586
Lymphopenia (Blood and lymphatic system disorders) | 33 | 27 | 32
Hemoglobin (Blood and lymphatic system disorders) | 587 | 574 | 572
Palpitations (Cardiac disorders) | 31 | 22 | 30
Hypertension (Cardiac disorders) | 90 | 149 | 206
Hypotension (Cardiac disorders) | 25 | 25 | 33
Sweating (General disorders) | 36 | 37 | 31
Weight Gain (General disorders) | 117 | 106 | 103
Fever (General disorders) | 61 | 48 | 74
Weight Loss (General disorders) | 76 | 80 | 101
Rigors/Chills (General disorders) | 36 | 35 | 43
Fatigue (General disorders) | 515 | 517 | 532
Insomnia (General disorders) | 125 | 136 | 134
Nail Changes (Skin and subcutaneous tissue disorders) | 20 | 29 | 42
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 452 | 459 | 444
Bruising (Skin and subcutaneous tissue disorders) | 31 | 31 | 36
Rash (Skin and subcutaneous tissue disorders) | 127 | 123 | 148
Dry Skin (Skin and subcutaneous tissue disorders) | 35 | 33 | 36
Pruritus (Skin and subcutaneous tissue disorders) | 57 | 59 | 66
Flushing (Skin and subcutaneous tissue disorders) | 35 | 33 | 31
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 37 | 27 | 33
Hot Flashes (Endocrine disorders) | 100 | 70 | 97
Heartburn (Gastrointestinal disorders) | 71 | 76 | 90
Distention (Gastrointestinal disorders) | 53 | 38 | 36
Taste Alteration (Gastrointestinal disorders) | 75 | 70 | 75
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 58 | 65 | 103
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 57 | 86 | 97
Vomiting (Gastrointestinal disorders) | 221 | 216 | 236
Anorexia (Gastrointestinal disorders) | 184 | 202 | 202
Dehydration (Gastrointestinal disorders) | 38 | 62 | 52
Constipation (Gastrointestinal disorders) | 377 | 351 | 355
Nausea (Gastrointestinal disorders) | 388 | 399 | 403
Diarrhea (Gastrointestinal disorders) | 240 | 265 | 260
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 60 | 181 | 188
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 38 | 40 | 42
Edema: Limb (Blood and lymphatic system disorders) | 115 | 82 | 89
Ast (Metabolism and nutrition disorders) | 75 | 63 | 86
Proteinuria (Metabolism and nutrition disorders) | 40 | 33 | 59
Creatinine (Metabolism and nutrition disorders) | 36 | 36 | 53
Hypoalbuminemia (Metabolism and nutrition disorders) | 62 | 71 | 79
Alt (Metabolism and nutrition disorders) | 78 | 66 | 76
Alkaline Phosphatase (Metabolism and nutrition disorders) | 74 | 64 | 83
Hyponatremia (Metabolism and nutrition disorders) | 77 | 75 | 98
Hypocalcemia (Metabolism and nutrition disorders) | 62 | 58 | 65
Hyperkalemia (Metabolism and nutrition disorders) | 35 | 32 | 42
Hyperglycemia (Metabolism and nutrition disorders) | 162 | 152 | 159
Hypokalemia (Metabolism and nutrition disorders) | 103 | 94 | 87
Hypoglycemia (Metabolism and nutrition disorders) | 29 | 31 | 42
Hypercalcemia (Metabolism and nutrition disorders) | 28 | 33 | 29
Hypomagnesemia (Metabolism and nutrition disorders) | 95 | 104 | 104
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 45 | 55 | 59
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 26 | 31 | 42
Mood Alteration - Depression (Nervous system disorders) | 80 | 90 | 101
Mood Alteration - Anxiety (Nervous system disorders) | 99 | 92 | 96
Memory Impairment (Nervous system disorders) | 27 | 32 | 29
Dizziness (Nervous system disorders) | 104 | 108 | 140
Neuropathy-Sensory (Nervous system disorders) | 435 | 432 | 434
Neuropathy-Motor (Nervous system disorders) | 57 | 39 | 48
Blurred Vision (Eye disorders) | 72 | 72 | 94
Pain - Other (General disorders) | 40 | 41 | 43
Pain: Chest /Thorax Nos (General disorders) | 32 | 34 | 30
Pain: Head/Headache (General disorders) | 128 | 142 | 193
Pain: Extremity-Limb (General disorders) | 93 | 101 | 142
Pain: Back (General disorders) | 99 | 109 | 127
Pain: Joint (General disorders) | 214 | 199 | 245
Pain: Bone (General disorders) | 61 | 52 | 58
Pain: Abdominal Pain Nos (General disorders) | 257 | 247 | 249
Pain: Muscle (General disorders) | 152 | 155 | 169
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 26 | 46 | 65
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 10 | 58 | 73
Cough (Respiratory, thoracic and mediastinal disorders) | 112 | 115 | 143
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 151 | 180 | 179
Incontinence, Urinary (Renal and urinary disorders) | 35 | 36 | 22
Urinary Frequency (Renal and urinary disorders) | 39 | 46 | 48

LIMITATIONS AND CAVEATS:
The results for both Overall Survival (OS) and Progression Free Survival (PFS) were based on the analysis performed on a data set frozen on August 26, 2011.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less